CLINICAL TRIAL: NCT04053478
Title: Effects of Ephedrine, Phenylephrine, Norepinephrine and Vasopressin on Contractility of Human Myometrium and Umbilical Vessels: An In-vitro Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-04
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Hypotension
Keywords: vasopressor; ephedrine; phenylephrine; norepinephrine; umbilical arteries; uterine contraction; fetal acidosis; vasopressin
MeSH Terms: conditions — Hypotension; Diabetes Insipidus | interventions — Ephedrine; Phenylephrine; Norepinephrine; Vasopressins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Myometrium + Ephedrine (Experimental): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of ephedrine
  Interventions: Drug: Ephedrine
- Myometrium + Phenylephrine (Experimental): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of phenylephrine
  Interventions: Drug: Phenylephrine
- Myometrium + Norepinephrine (Experimental): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of norepinephrine
  Interventions: Drug: Norepinephrine
- Myometrium + Vasopressin (Experimental): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of vasopressin
  Interventions: Drug: Vasopressin
- Umbilical artery + Ephedrine (Experimental): The umbilical artery samples are bathed in physiological salt solution (PSS) with increasing concentrations of ephedrine
  Interventions: Drug: Ephedrine
- Umbilical artery + Phenylephrine (Experimental): The umbilical artery samples are bathed in physiological salt solution (PSS) with increasing concentrations of phenylephrine
  Interventions: Drug: Phenylephrine
- Umbilical artery + Norepinephrine (Experimental): The umbilical artery samples are bathed in physiological salt solution (PSS) with increasing concentrations of norepinephrine
  Interventions: Drug: Norepinephrine
- Umbilical artery + Vasopressin (Experimental): The umbilical artery samples are bathed in physiological salt solution (PSS) with increasing concentrations of vasopressin
  Interventions: Drug: Vasopressin
- Umbilical vein + Ephedrine (Experimental): The umbilical vein samples are bathed in physiological salt solution (PSS) with increasing concentrations of ephedrine
  Interventions: Drug: Ephedrine
- Umbilical vein + Phenylephrine (Experimental): The umbilical vein samples are bathed in physiological salt solution (PSS) with increasing concentrations of phenylephrine
  Interventions: Drug: Phenylephrine
- Umbilical vein + Norepinephrine (Experimental): The umbilical vein samples are bathed in physiological salt solution (PSS) with increasing concentrations of norepinephrine
  Interventions: Drug: Norepinephrine
- Umbilical vein + Vasopressin (Experimental): The umbilical vein samples are bathed in physiological salt solution (PSS) with increasing concentrations of vasopressin
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Ephedrine — Ephedrine in solution, at applicable concentrations based on literature
  Arms: Myometrium + Ephedrine; Umbilical artery + Ephedrine; Umbilical vein + Ephedrine
Drug: Phenylephrine — Phenylephrine, at applicable concentrations based on literature
  Arms: Myometrium + Phenylephrine; Umbilical artery + Phenylephrine; Umbilical vein + Phenylephrine
Drug: Norepinephrine — Norepinephrine, at applicable concentrations based on literature
  Arms: Myometrium + Norepinephrine; Umbilical artery + Norepinephrine; Umbilical vein + Norepinephrine
Drug: Vasopressin — Vasopressin, at applicable concentrations based on literature
  Arms: Myometrium + Vasopressin; Umbilical artery + Vasopressin; Umbilical vein + Vasopressin

SUMMARY:
Hypotension is one of the most common adverse effects of spinal anesthesia for cesarean deliveries, affecting as many as 55-90% of mothers. Hypotension during cesarean deliveries can have detrimental effects on the mother and neonate. Various vasopressors, such as ephedrine, phenylephrine and more recently norepinephrine, have been used for the prevention and treatment of hypotension at cesarean deliveries.

Ephedrine was historically considered as the gold standard vasopressor for the management of hypotension during cesarean deliveries. This was based on studies in animal models that showed preserved uteroplacental circulation with ephedrine and not with phenylephrine. However, multiple studies in the past several decades have shown that phenylephrine compared with ephedrine results in a more favorable fetal acid-base status. Consequently, the use of phenylephrine for blood pressure management during cesarean deliveries increased. Recently, norepinephrine was introduced in the obstetrical practice for the management of hypotension at cesarean deliveries, due to its ability to maintain maternal cardiac output better than phenylephrine.

Studies have also investigated the use of vasopressin to limit hypotension during CD. There have been case reports of successful vasopressin usage to treat post-spinal hypotension after CD in patients with advanced idiopathic pulmonary arterial hypertension as well as severe mitral stenosis with pulmonary hypertension. Its effect was associated with hemodynamic stability without evidence of harm to the mother or child. However, much controversy still exists surrounding the choice of vasopressor in the obstetric population, in large part due to their varying efficacies, and maternal and fetal effects.

Vasopressors used for the treatment of hypotension during cesarean deliveries can have significant direct or indirect effects on the perfusion of uteroplacental and umbilical vessels. Reduction of uteroplacental perfusion and constriction of umbilical vessels can result in fetal acidosis, however, the mechanisms for these effects are unclear. The investigators hypothesize that ephedrine, phenylephrine and norepinephrine and vasopressin have variable effects on the contractility of pregnant myometrium and umbilical arteries due to their variable actions on adrenergic alpha (α) and beta (β) receptors, as well as vasopressin1 and vasopressin2 receptors located in these tissues.

DETAILED DESCRIPTION:
One of the major concerns addressed in the literature is the risk of fetal acidosis related to the use of vasopressors, which varies according to the type of drug used. Since severe fetal acidosis is associated with a two- and four-fold increase in neonatal morbidity and mortality, respectively, it is important to understand the mechanism by which these medications may contribute to fetal acidosis.

It is well known that reduced uteroplacental blood flow can result in impaired fetal oxygenation and fetal acidosis. This can occur indirectly via compression of vessels due to myometrial contractions or directly by vasoactive effects on umbilical vessels. So far, no studies have directly explored the role of the aforementioned vasopressors on myometrial contractions and umbilical vessel vasoconstriction. An in-vitro approach in isolated tissues will eliminate many clinical confounding variables, allowing direct comparison of the drugs in a controlled environment, and providing insight into the contractile mechanisms responsible for their neonatal effects.

There is currently no consensus as to which vasopressor is best for the management of hypotension in obstetric patients and the mitigation of fetal acidosis. A survey of the members of the Society of Obstetric Anesthesia and Perinatology suggested significant variation in the practice of vasopressor use during cesarean deliveries. The evidence from animal studies contradicts the effects seen in human studies. This is possibly related to species differences in adrenergic receptor distribution, affinity to vasopressors, or placental transfer of vasopressors. It is well known that reduced uteroplacental blood flow can result in impaired fetal oxygenation and fetal acidosis. This can occur indirectly via compression of vessels due to myometrial contractions or directly by vasoactive effects on umbilical arteries. However, none of the studies so far have directly explored the role of the aforementioned vasopressors on myometrial contractions and umbilical artery vasoconstriction. An in-vitro approach in isolated tissues will eliminate many clinical confounding variables, allowing direct comparison of the drugs in a controlled environment, and providing insight into the contractile mechanisms responsible for their neonatal effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Patients of 19-40 years
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring elective primary or first repeat caesarean delivery
* Patients undergoing caesarean delivery under spinal anesthesia

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients in labor and those receiving oxytocin for induction of labor
* Emergency caesarean delivery in labor
* Patients who have had previous uterine surgery or >1 previous caesarean delivery
* Patients with any condition predisposing to uterine atony
* Patients on medications that could affect myometrial contractility, such as insulin, nifedipine, labetolol or magnesium sulfate.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Motility index | 4 hours
  Motility index (MI) is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  Frequency and amplitude are secondary outcome measures as described below.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 4 hours
  The maximum extent of uterine muscle and umbilical vessel contractions, measured in grams (g). The analysis is undertaken by attaching myometrial strips and umbilical vessel rings between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 4 hours
  The number of contractions in uterine muscle (myometrium) and umbilical vessel rings over 10 minutes, spontaneously and in response to an agonist.
  The analysis is undertaken by attaching myometrial strips and umbilical vessel rings between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No